CLINICAL TRIAL: NCT00805519
Title: Efficacy and Safety of Prednisolone and Chloroquine Add on Therapy in Osteoarthritis of the Knee Treated With Fixed Dose Combination of Glucosamine and Chondroitin Sulfate.
Brief Title: Efficacy and Safety of Prednisolone and Chloroquine Add on Therapy in Osteoarthritis of the Knee
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ardabil University of Medical Sciences (Other)
Responsible Party: Shahab Bohlooli, Pharmacology Dept., Faculty of Medicine, ArdabilUMS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 870919
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Last update posted 2010-04-30 (Estimated); Status verified 2010-04

CONDITIONS: Osteoarthritis of the Knee
Keywords: Osteoarthritis of the Knee; Glucosamine Chondroitin sulfate; Prednisolone; Chloroquine
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Glucosamine; Chondroitin Sulfates; Prednisolone; Chloroquine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Glucosamine and chondroitin sulfate (Active Comparator): in this group patients will receive Glucosamine and chondroitin sulfate oral dietary supplementation
  Interventions: Drug: Glucosamine and chondroitin sulfate
- P :glucosa, chondroitin, Prednis (Experimental): in this group patients will receive glucosamine and chondroitin sulfate plus Prednisolone oral administration
  Interventions: Drug: glucosamine and chondroitin sulfate plus Prednisolone
- Glucosa, Chondroitin, Chloroquine (Experimental): in this group pateints will orally receive Glucosamine and Chondroitin sulfate plus Chloroquine.
  Interventions: Drug: Glucosamine and Chondroitin sulfate plus Chloroquine
- Glucosa, Chondro, Prednis,Chloroq (Experimental): in this group patients will receive Glucosamine and Chondroitin sulfate plus Prednisolone and Chloroquine
  Interventions: Drug: Glucosamine,Chondroitin sulfate,Prednisolone,Chloroquine

INTERVENTIONS:
Drug: Glucosamine and chondroitin sulfate — In this arm fixed dose glucosamine (400 mg) and chondroitin sulfate (500 mg)combination will be administrated to the patients, daily.
  Arms: Glucosamine and chondroitin sulfate
Drug: glucosamine and chondroitin sulfate plus Prednisolone — In this arm fixed dose glucosamine (400 mg) and chondroitin sulfate (500 mg)combination will be administrated to the patients as baseline therapy, daily. also,the patients will receive Prednisolone 5 mg/day
  Arms: P :glucosa, chondroitin, Prednis
Drug: Glucosamine and Chondroitin sulfate plus Chloroquine — In this arm fixed dose glucosamine (400 mg) and chondroitin sulfate (500 mg)combination will be administrated to the patients as baseline therapy, daily. also,the patients will receive chloroquine 150 mg every two days.
  Arms: Glucosa, Chondroitin, Chloroquine
Drug: Glucosamine,Chondroitin sulfate,Prednisolone,Chloroquine — In this arm fixed dose glucosamine (400 mg) and chondroitin sulfate (500 mg)combination will be administrated to the patients as baseline therapy, daily. also,the patients will receive prednisolone 5 mg/day and chloroquine 150 mg every two days.
  Arms: Glucosa, Chondro, Prednis,Chloroq

SUMMARY:
This study was conducted to evaluate the efficacy and safety of prednisolone and chloroquine add on therapies to combined glucosamine, chondroitin sulfate in osteoarthritis of the knee which will be done in contrast to combined glucosamine sulfate and chondroitin.

DETAILED DESCRIPTION:
Fixed dose glucosamine, chondroitin sulfate combination is a treatment to osteoarthritis with some controversy about efficacy. it seems that addition of other agents may improve efficacy and decrease the required dose and cost. common oral corticosteroids such as low dose prednisolone and chloroquine are candidate for such add on therapies. nevertheless, add on therapy may expose the patients to new side effects which should followed and addressed.

In this investigator blinded controlled trial, 240 patients with diagnosed osteoarthritis of knee will be enrolled to the study. the patients will randomly be assigned to one of four groups of G (glucosamine and chondroitin sulfate ), P (Glucosamine and Chondroitin sulfate plus Prednisolone), C (Glucosamine and Chondroitin sulfate plus Chloroquine) and PC (Glucosamine and Chondroitin sulfate plus Prednisolone and Chloroquine). each group will consist 60 patients. the investigator(s) will be blind to the groups and interventions.

ELIGIBILITY:
Inclusion Criteria:

* men and non-pregnant women, age 40-85 years with primary OA of at least one knee.

Exclusion Criteria:

* secondary arthritis related to systemic inflammatory arthritis (including rheumatoid arthritis, psoriatic arthritis, post-infectious arthritis and metabolic arthritis, traumatic arthritis or surgical joint replacement)corticosteroid use:

  * oral corticosteroid within the previous 14 days
  * intramuscular corticosteroid within 30 days
  * intraarticular corticosteroid into the study knee within 90 days
  * intra-articular corticosteroid into any other joint within 30 days or
  * topical corticosteroid at the site of application within 14 days
* ongoing use of prohibited medication including NSAID, other oral analgesic, muscle relaxant, or low-dose antidepressant for any chronic pain management
* glucosamine or chondroitin within the previous six months
* history of alcohol or drug abuse
* lactation
* concomitant skin disease at the application site
* current application for disability benefits on the basis of knee osteoarthritis; fibromyalgia; other painful or disabling condition affecting the knee

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2009-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome measures is defined as the change from baseline to final assessment of the study knee in the 3 core continuous variables pain and physical function, assessing using the WOMAC subscales, and patient global assessment (PGA) | Baseline
The primary outcome measures is defined as the change from baseline to final assessment of the study knee in the 3 core continuous variables pain and physical function, assessing using the WOMAC subscales, and patient global assessment (PGA) | the outcome is assessed at 6 weeks after baseline visit
The primary outcome measures is defined as the change from baseline to final assessment of the study knee in the 3 core continuous variables pain and physical function, assessing using the WOMAC subscales, and patient global assessment (PGA) | the outcome is assessed at 12 weeks after baseline visit

SECONDARY OUTCOMES:
The secondary measure will be changes in stiffness | the outcome is assessed at baseline visit
The secondary measure will be changes in stiffness | the outcome is assessed at 6 weeks after baseline visit
The secondary measure will be changes in stiffness | the outcome is assessed at 12 weeks after baseline visit

CONTACTS AND LOCATIONS:
Overall Officials: Shahab Bohlooli, PhD, Principal Investigator — Pharmacology Dept, Faculty of Medicine, ArdabilUMS; Marina Jastan, MD, Principal Investigator — Rheomatology clinic, Faculty of Medicine, ArdabilUMS
Locations (1):
- ArdabiUMS Clinic of Rheumatology, Ardabil, Ardabil Province, Iran